CLINICAL TRIAL: NCT01378988
Title: A Phase II, Randomized, Open-Label, Single Center, Pharmacokinetic and Pharmacodynamic Study of Dexmedetomidine in Pediatric Subjects Aged 12 Months Through <24 Months
Brief Title: Phase II Pharmacokinetic and Pharmacodynamic Study of DEX in Subjects Aged 12 Months Through <24 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX-11-01
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-06

CONDITIONS: Sedation; Pain
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose level 1 (Experimental): Dexmedetomidine 0.7 mcg/kg loading dose and 0.5 mcg/kg/hr maintenance infusion
  Interventions: Drug: Dexmedetomidine
- Dose level 2 (Experimental): Dexmedetomidine 1.0 mcg/kg loading dose and 0.75 mcg/kg/hr maintenance infusion
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — For sedation according to protocol

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic, pharmacodynamic, and safety of dexmedetomidine at 2 different dose levels in pediatric subjects, aged 12 months through <24 months, administered as an intravenous loading dose followed by continuous infusion for a minimum of 6 hours and up to 24 hours in an intensive care setting.

DETAILED DESCRIPTION:
Phase II, randomized, open-label, single-center, study evaluating the pharmacokinetics and pharmacodynamics of dexmedetomidine in pediatric subjects across two dose levels (Dose Level 1 consists of a 0.7 mcg/kg loading dose immediately followed by a 0.5 mcg/kg/hr maintenance infusion; Dose Level 2 consists of a 1.0 mcg/kg loading dose immediately followed by a 0.75 mcg/kg/hr maintenance infusion). The study population will consist of intubated and mechanically ventilated pediatric subjects who require sedation in an intensive care setting for a minimum of 6 hours but not to exceed 24 hours. Subjects eligible for enrollment are 12 months to <24 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 12 months to <24 months of age at screening.
2. Subject is intubated and mechanically ventilated in an intensive care setting and is anticipated to require a minimum of 6 hours of continuous IV sedation.
3. Subject has adequate renal function, defined as: Serum creatinine ≤1.0 mg/dL.
4. The subject's parent(s) or legal guardian(s) must voluntarily sign and date the informed consent document approved by the Institutional Review Board.

Exclusion Criteria:

1. Pediatric subjects with neurological conditions that prohibit an evaluation of sedation such as:

   * Diminished consciousness from increased intracranial pressure
   * Extensive brain surgery (surgery requiring intracranial pressure monitor)
   * Diminished cognitive function per Principal Investigator (PI) discretion
   * Subjects with immobility from neuromuscular disease or continuous infusion of neuromuscular blocking agents.
2. Subjects with second degree or third degree heart block unless subject has a permanent pacemaker or pacing wires are in situ.
3. Subjects who have hepatic impairment as defined by a serum glutamic-pyruvic transaminase/alanine aminotransferase (SGPT/ALT) >90 U/L at the time of screening.
4. Subjects who have hypotension, based on repeat assessments within 15 minutes preceding the start of study drug, defined as: Systolic blood pressure (SBP) <70 mmHg.
5. Pre-existing bradycardia based on repeated assessments within 15 minutes preceding the start of study drug, defined as: Heart rate (HR) <70 bpm.
6. Subject who have acute thermal burns involving more than 15 percent total body surface area.
7. Subjects who have a known allergy to dexmedetomidine, midazolam or fentanyl.
8. Subject who has received dexmedetomidine within 15 hours prior to the start of study drug.
9. Subjects with a life expectancy that is <72 hours.
10. Subjects that are expected to have hemodialysis (continuous hemofiltration), peritoneal dialysis or extracorporeal membrane oxygenation (ECMO) treatments within 48 hours prior to the start of study drug or during the duration of the study.
11. Subjects who have been treated with α-2 agonists/antagonists within 2 weeks.
12. Subjects with a spinal cord injury above T5 (5th Thoracic Vertebra).
13. Subjects who have received another investigational drug as part of an investigational drug study within the past 30 days.
14. Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of this clinical study.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Chrysostomou, MD, Principal Investigator — Children's Hospital of Pittusburgh of UPMC
Locations (1):
- Children's Hospital of Pittusburgh of UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Evaluable Population consisted of all subjects who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.43 (0.312) | 1.45 (0.274) | 1.44 (0.249)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC0-∞)
Description: Area under the plasma concentration-time curve of dexmedetomidine at 0 to Infinity hours
Time Frame: 30 minutes prior to loading dose (LD); 5 minutes before finishing LD; 0.5, 1, 2 and 4-6 hours during maintenance infusion (MI); 30 minutes prior (within 24 hours of start of MI) and 10 minutes, 0.5, 1, 2, 4 and 10 hours end of MI
Population: Full Evaluable Population consisted of all subjects who received study drug for at least 5 hours with adequate PK samples to estimate primary parameters.
Measure: Mean (Standard Deviation); unit: picogram*hour per millilitre
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
picogram*hour per millilitre | 4639.17 (4058.1893) | 14203.544 (13051.6850)

2. Primary Outcome: Observed Peak Plasma Concentration (Cmax)
Description: Maximum observed concentration of dexmedetomidine in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picogram per millilitre
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
picogram per millilitre | 4499.925 (5826.7367) | 11737.387 (3549.7923)

3. Primary Outcome: Steady State Concentration (Css)
Description: Concentration of dexmedetomidine at steady state in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picogram per millilitre
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
picogram per millilitre | 752.298 (658.0848) | 2303.277 (2116.4895)

4. Primary Outcome: Terminal Elimination Half-life (t1/2)
Description: Terminal elimination half-life of dexmedetomidine. Half-life is the time required for plasma concentration of the drug to decrease by 50%.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
Hours | 1.958 (0.3765) | 2.260 (1.2205)

5. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Observed time to reach maximum plasma concentration of dexmedetomidine, expressed in hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
Hours | 0.083 (0.0) | 0.283 (0.3464)

6. Primary Outcome: Weight-Adjusted Plasma Clearance (CLw)
Description: Weight-Adjusted Plasma Clearance of dexmedetomidine after intravenous administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre per Hours per Kilogram
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
Litre per Hours per Kilogram | 1.292 (1.1300) | 0.617 (0.3815)

7. Primary Outcome: Plasma Clearance (CL)
Description: Clearance of dexmedetomidine after intravenous administration. Clearance is the rate at which the drug is removed from the plasma after the dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre per Hour
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
Litre per Hour | 12.192 (9.5770) | 5.836 (2.9357)

8. Primary Outcome: Volume of Distribution (Vd)
Description: Volume of distribution of dexmedetomidine after intravenous administration. Volume of distribution measures how much the drug spreads through the body after the dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
Litre | 31.845 (20.4351) | 15.780 (3.5461)

9. Primary Outcome: Weight-Adjusted Volume of Distribution (Vdw)
Description: Weight-Adjusted Volume of distribution of dexmedetomidine after intravenous administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre per Kilogram
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
Litre per Kilogram | 3.343 (2.4910) | 1.590 (0.6201)

10. Primary Outcome: Average Total Faces, Legs, Activity, Cry, and Consolability (FLACC) Score
Description: FLACC scale is a 5 category observational measure to assess pediatric pain on face, legs, activity, cry and consolability. Responses in each category are scored between 0 to 2 (0 = normal, relaxed to 2 = upset, rigid), for a maximum total score of 10.
Time Frame: Prior to loading dose and every hour during the maintenance infusion; within 5 minutes after any fentanyl administration during DEX infusion or every 4 hours in case of continuous fentanyl infusion; within 5 minutes prior and after titration of fentanyl
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
units on a scale | 1.575 (2.2274) | 3.220 (2.1707)

11. Primary Outcome: Absolute Time That Subject is in UMSS Range 2-4 During Treatment Period
Description: The level of sedation will be assessed using the University of Michigan Sedation Scale (UMSS).
  Score 0 (awake/alert); Score 1 (sleepy/responds appropriately); Score 2 (somnolent/arouses to light stimuli); Score 3 (deep sleep/arouses to deeper physical stimuli); Score 4 (unarousable).
  The UMSS scores obtained just prior the loading dose (LD) and 5 and 10 minutes during LD; 0, 5, 10, 15, 30, and 60 minutes and thereafter every 4 hours of the maintenance infusion; within 5 minutes of obtaining each pharmacokinetic sample; within 5 minutes prior and after any midazolam rescue during dexmedetomidine infusion period.
Time Frame: During the treatment (6 to 24 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
Hours | 3.6 (3.48) | 5.8 (0.38)

12. Primary Outcome: Number of Subjects Who Received Rescue Medication for Sedation and Analgesic
Description: Participants who received rescue medication midazolam for sedation and/or fentanyl for analgesic during study drug Infusion
Time Frame: During the treatment (6 to 24 hours)
Population: Full Evaluable Population consisted of all subjects who received study drug for at least 5 hours with adequate pharmacokinetic samples to estimate primary parameters.
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 3
participants
  Midazolam for sedation | 1 | 1
  Fentanyl for Analgesic | 1 | 2

ADVERSE EVENTS:
Groups:
- Dose Level 1: Dexmedetomidine 0.7 mcg/kg loading dose and 0.5 mcg/kg/hr maintenance dose
- Dose Level 2: Dexmedetomidine 1.0 mcg/kg loading dose and 0.75 mcg/kg/hr maintenance dose
Arm/Group | Dose Level 1 | Dose Level 2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=2) | Dose Level 2 (N=3)
Pyrexia (General disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No